CLINICAL TRIAL: NCT02652923
Title: Contrast Ultrasound Detection of Sentinel Lymph Nodes in Breast Cancer Patients
Brief Title: Contrast Ultrasound Detection of Sentinel Lymph Nodes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); GE Healthcare (Industry); Siemens Medical Solutions (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 15P.487; R01CA172336 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-01-12 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: ultrasound contrast agent; lymphosonography; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sonazoid; perfluorobutane; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1 - volunteers (Experimental): Subdermal low (1.0 ml) or high (2.0 ml) dose injection of the ultrasound contrast agent Sonazoid divided into four individual aliquots at four locations (12, 3, 6, and 9 o'clock) around a 2 cm in diameter region in the mid-upper outer quadrant of the left breast, followed a week later by the other dose injected in the same fashion into the right breast.
  Interventions: Drug: Sonazoid; Perflubutane for Injection
- Part 2 - patients (Experimental): Subdermal injection of the ultrasound contrast agent of Sonazoid divided into four individual aliquots at four locations (12, 3, 6, and 9 o'clock) around the breast cancer. Subjects will receive an injection of either a low (1.0 ml) or a high (2.0 ml) dose of Sonazoid depending on the outcome of the Part 1 safety and tolerability study.
  Interventions: Drug: Sonazoid; Perflubutane for Injection

INTERVENTIONS:
Drug: Sonazoid; Perflubutane for Injection — subdermal injection into the breast of Sonazoid (1 or 2 ml) divided into four individual aliquots at four locations (12, 3, 6, and 9 o'clock)
  Other Names: ultrasound microbubble contrast agent

SUMMARY:
This is a two part, open label, non-randomized trial of women with a breast cancer diagnosis scheduled for excisional surgery and sentinel lymph node (SLN) evaluation.

Part 1 is a two-period, crossover, dose-finding study, which will be performed in 12 healthy female volunteers to determine the optimal dose as well as the safety and tolerability of the tissue-specific, contrast agent Sonazoid (GE Healthcare, Oslo, Norway) for human lymphatic applications. In Part 2 lymphosonographic SLN identification will be compared to that of isotope mapping during surgery on 90 female, breast cancer patients.

DETAILED DESCRIPTION:
This is a two part, open-label, non-randomized trial that will be conducted at Thomas Jefferson University (TJU). Initially in Part 1, a two-period, crossover, dose-finding study will be performed in 12 healthy female volunteers to determine the optimal dose as well as the safety and tolerability of the tissue-specific, contrast agent Sonazoid (GE Healthcare, Oslo, Norway) for human lymphatic applications. Each volunteer will receive an injection of a low or a high dose in a blinded, sequence-randomized allocation schedule. Screening and baseline assessments/procedures will be obtained. Each volunteer will receive their subdermal, low or high dose of Sonazoid divided into four individual aliquots at four locations (12, 3, 6, and 9 o'clock) around a 2 cm in diameter region in the mid-upper outer quadrant of the left breast.

Contrast enhanced ultrasound imaging (CEUS) will be performed immediately after Sonazoid administration (i.e., lymphosonography) to identify the number, location and course of the lymphatic channels (LCs) and SLNs using a S3000 scanner (Siemens Medical Solutions, Mountain View, CA) with a high frequency, broad bandwidth linear array. CEUS evaluations will be repeated at 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours and 24 hours post Sonazoid administration. The safety and tolerability of Sonazoid will be closely monitored throughout this safety and tolerability, dose-finding study.

Following at least a one week of washout, the upper outer quadrant of the right breast will be injected with the alternate dose of Sonazoid and lymphosonography will again be used to identify the number, location and course of the LCs and SLNs. Volunteers who received the low dose during their first visit will receive the high dose the next time around and vice versa in a 1:1 ratio. All procedures from the initial visit will be repeated (see above), except that the left breast (injected initially) will be assessed sonographically for the presence of contrast-enhanced tissues (injection site as well as lymphatic structures) prior to contrast administration in the right breast.

In Part 2 lymphosonography will compare SLN identification to that of isotope mapping during surgery on 90 female, breast cancer patients. A state-of-the-art S3000 scanner with contrast-specific imaging capabilities will be used to localize lymphatic drainage from breast cancers after subdermal administration of Sonazoid. The number and locations of the SLNs identified by the two imaging modalities (CEUS and isotope mapping) will be compared with dye-guided surgery as the reference standard for SLN detection. Moreover, as each SLN is resected it will be assessed ex vivo for the presence of radioactivity (using a gamma probe), Sonazoid (using CEUS) and blue dye (via visual inspection by the surgeon). All SLNs that are surgically removed will be documented and sent for histopathologic evaluation.

Trial Population: Part 1 will consist of 12 healthy, adult female volunteers in the initial safety, tolerability and dosing study.

In Part 2, 90 adult women, who have breast cancer and are scheduled for a surgical excision and SLN evaluation, will be enrolled in a clinical trial at TJU.

Statistical Methodology: Our statistical analysis will address four major questions:

* Is subdermal administration of Sonazoid in humans safe and tolerable?
* Can an optimal and efficacious dose of Sonazoid for lymphosonography be established?
* Does lymphosonography identify more SLNs in patients with breast cancer than isotope mapping (with Tc-99m sulfur colloids)?
* Does lymphosonography identify more SLNs with metastatic deposits in patients with breast cancer compared to isotope mapping?

ELIGIBILITY:
Inclusion Criteria:

* Part 1:

  * Be female.
  * Be at least 21 years of age.
  * Must have a body mass index (BMI) greater or equal to 19 and less than or equal to 33.
  * Be able to comprehend the full nature, purpose and risks of the study.
* Part 2:

  * Be female.
  * Be diagnosed with breast cancer.
  * Be scheduled for a surgical excision with SLN evaluation.
  * Be at least 21 years of age.
  * Be medically stable.
  * If of child-bearing potential, must have a negative pregnancy test.
  * Be able to comply with study procedures.
  * Have read and signed the IRB-approved Informed Consent form for participating in the study.

Exclusion Criteria:

* Part 1:

  * A history of chest wall trauma or surgery, or dermatologic disorders, which could be expected to disrupt lymphatic drainage of the chest wall.
  * A history of surgical breast augmentation, reduction, or biopsy.
  * Lymphedema or chronic edema.
  * Females who are pregnant or nursing or are actively lactating.
  * Exposure to ultrasound contrast agents in the 1 month prior to study initiation.
  * Known hypersensitivity to ultrasound contrast agents.
  * Patients with a history of anaphylactic allergy to eggs or egg products, manifested by one or more of the following symptoms: generalized urticaria, difficulty in breathing, swelling of the mouth and throat, hypotension, or shock.
  * Significant axillary, supraclavicular, or other chest wall palpable adenopathy.
  * Evidence of current ongoing illicit drug use or average alcohol use of greater than 2 drinks a day.
  * Use of more than 5 cigarettes/day.
  * Participation in an investigational drug study within the period starting 1 month before study drug administration.
  * Subject is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder within the last 5 years. Subjects who have had situational depression may be enrolled in the study at the discretion of the Investigator.
  * Subject has a history of any illness that, in the opinion of the study Investigator, might confound the results of the study or poses an additional risk to the subject by his participation in the study.
  * An estimated creatinine clearance of ≤80 ml/min based on the Cockcroft-Gault equation. An actual creatinine clearance, as determined by a 24 hour urine collection, may be used in place of the Cockcroft-Gault equation. Subjects who have an actual or estimated creatinine clearance 70 ml/min may be enrolled at the discretion of the investigator.
  * A history of neoplastic disease, with the exception of non-melanoma skin cancer.
  * Any other condition precluding subject participation as per investigator judgment.
* Part 2:

  * Females who are pregnant or nursing.
  * Patients who have had prior breast reduction.
  * Patients with a prior axillary procedure on the side scheduled for SLN evaluation.
  * Patients with other primary cancers requiring systemic treatment.
  * Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable. For example:
  * Patients on life support or in a critical care unit.
  * Patients with unstable occlusive disease (e.g., crescendo angina)
  * Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia.
  * Patients with uncontrolled congestive heart failure (NYHA Class IV)
  * Patients with recent cerebral hemorrhage.
  * Patients who have undergone surgery within 24 hours prior to the study sonographic examination.
  * Patients with a history of anaphylactic allergy to eggs or egg products, manifested by one or more of the following symptoms: generalized urticaria, difficulty in breathing, swelling of the mouth and throat, hypotension, or shock. (Subjects with nonanaphylactic allergies to eggs or egg products may be enrolled in the study, but must be watched carefully for 1 h following the administration of Sonazoid).
  * Patients with cardiac shunts or unstable cardiopulmonary conditions.
  * Patients with congenital heart defects.
  * Patients with severe emphysema, pulmonary vasculitis, pulmonary hypertension or a history of pulmonary emboli.
  * Patients who have received any contrast medium (X-ray, MRI, CT or US) in the 24 hours prior to the research US exam
  * Patients with respiratory distress syndrome.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Dose optimization (1.0 vs 2.0 ml) based on the degree and duration of Sonazoid contrast-enhancement of the visualized LCs and SLNs | Up to 4 months
  To establish, in healthy, female volunteers, the optimal dose of subdermaly administrated Sonazoid (an ultrasound contrast agent) employed for contrast enhanced ultrasound imaging (CEUS)
Number of subdermal Sonazoid volunteers with AEs, clinical assessments, and safety laboratory tests outside normal ranges (established by historical controls) | Up to 4 months
  To assess the safety and tolerability of subdermal administration of Sonazoid in 12 female, healthy volunteers.
Number SLNs in patients with breast cancer identified by lymphosonography and by isotope mapping with Tc-99m sulfur colloids. | Up to 34 months
  To determine if CEUS of subdermally administrated Sonazoid (i.e., lymphosonography) identify more sentinel lymph nodes (SLNs) in patients with breast cancer compared to isotope mapping (with Tc-99m sulfur colloids) using blue dye and surgical dissection as the reference standard. The fundamental hypothesis is that on average lymphosonography will detect 3.2 SLNs compared to 2.7 with isotope mapping.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Forsberg, PhD, Principal Investigator — Radiology; Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to the research community upon request after the completion of the study in accordance with NIH rules and regulations.